CLINICAL TRIAL: NCT06984510
Title: Accelerated Biological Aging is Associated With Increased Risk of T2DM in the MASLD Population: a Cohort Study
Brief Title: Accelerated Biological Aging is Associated With Increased Risk of T2DM in the MASLD Population
Status: Recruiting | Type: Observational
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-070RS-01; MR-33-25-026098 (Registry Identifier: medicalresearch.cn)
Record Dates: First submitted 2025-05-11; First posted 2025-05-22 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Metabolic Dysfunction-Associated Steatotic Liver Disease; Biological Age
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MASLD group: participants with MASLD at baseline
  Interventions: Other: Observational
- non-MASLD group: participants without MASLD at baseline
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational

SUMMARY:
The association between biological aging and type 2 diabetes mellitus (T2DM) incidence in individuals with and without metabolic dysfunction-associated steatotic liver disease (MASLD) remains unclear.We assessed biological age by calculating phenotypic age (PhenoAge), Klemera-Doubal method (KDMAge), and homeostatic dysregulation (HDAge). To examine the association of biological ageing with the risk of T2DM, cox regression models were conducted. Furthermore, we applied survival analysis, restricted cubic spline models and population attributable fraction (PAF) to further evaluate the association between biological ageing and T2DM incidence.

ELIGIBILITY:
Inclusion Criteria:

1. Abdominal ultrasound data available in annual health check-up records
2. At least one of the following five metabolic indicators recorded annually:

(1) Body mass index (BMI) or waist circumference (2) Blood pressure (3) Serum triglycerides (4) High-density lipoprotein cholesterol (HDL-C) (5) Fasting plasma glucose or glycated hemoglobin (HbA1c)

Exclusion Criteria:

1. Age <20 or >90 years
2. Other causes of hepatic steatosis (e.g., alcoholic liver disease or hepatitis B infection)
3. Type 2 diabetes mellitus at baseline
4. Missing baseline data for any of the following variables: systolic blood pressure, albumin, alkaline phosphatase, blood urea nitrogen, creatinine, glycated hemoglobin (HbA1c), total cholesterol, lymphocyte percentage, white blood cell count, mean corpuscular volume, uric acid, fasting plasma glucose, and red cell distribution width (RDW)

Ages: 20 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This retrospective cohort study is based on physical examination at the Physical Examination Center of The First Affiliated Hospital of Ningbo University and included participants aged 20 to 90 years. Individuals included had available abdominal ultrasound data and at least one recorded metabolic indicator per year. Participants with type 2 diabetes at baseline or with other causes of hepatic steatosis were excluded. The study population was categorized into MASLD and non-MASLD groups for comparative analysis.
Sampling Method: Non-Probability Sample
Enrollment: 2720 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of onset T2DM | through study completion, an average of 3 year

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Ningbo University Ningbo, Zhejiang, China, 315000, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No